CLINICAL TRIAL: NCT05131243
Title: the Role of ctDNA in Predicting the Recurrence Risk of Stage Ⅱ and Ⅲ Colorectal Cancer and the Dynamic Changes in ctDNA of Patients With Adjuvant Chemotherapy
Brief Title: the Role of ctDNA in Predicting the Recurrence Risk of Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FZ-CON-001
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer Stage II; Colorectal Cancer Stage III
Keywords: ctDNA; Adjuvant chemotherapy; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA positive patients (Experimental): Postoperative ctDNA-positive patients will receive chemotherapy for 6 months.The ctDNA dynamic detection and imaging examination will be completed every 3 months, and tumor markers will be detected in each chemotherapy cycle.
  Interventions: Procedure: Chemotherapy time
- ctDNA negative patients (Active Comparator): Postoperative ctDNA-negative patients will receive chemotherapy for 3 months. The ctDNA dynamic detection and imaging examination will be completed every 3 months, and tumor markers will be detected in each chemotherapy cycle.
  Interventions: Procedure: Chemotherapy time

INTERVENTIONS:
Procedure: Chemotherapy time — 6 months of chemotherapy
  Arms: ctDNA positive patients
Procedure: Chemotherapy time — 3 months of chemotherapy
  Arms: ctDNA negative patients

SUMMARY:
The purpose of this study was to observe the relationship between ctDNA as a molecular marker of colorectal cancer and the risk of postoperative recurrence.

DETAILED DESCRIPTION:
In this clinical study, ctDNA will be detected in postoperative patients with stage Ⅱ and Ⅲ colorectal cancer to evaluate the correlation between ctDNA and the risk of postoperative recurrence. According to the dynamic changes of ctDNA after adjuvant chemotherapy, the correlation between ctDNA and postoperative DFS will be compared, and the feasibility of ctDNA as a molecular marker to evaluate the risk of postoperative recurrence of colorectal cancer will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with colorectal cancer diagnosed pathologically as stage Ⅱ and stage Ⅲ.
* 2. The patient underwent radical surgical treatment.
* 3. The patient has the results of genetic genetic testing for gastrointestinal tumors, including the genetic mutation status of MMR genes and related genes (MLH1, MSH2, MSH6, PMS2, MLH3, EPCAM).
* 4. The patient understands and is willing to sign a written informed consent document.
* 5. During the treatment process, the patient can cooperate to provide samples of each node.
* 6. The patient can provide corresponding clinical materials, including but not limited to case diagnosis, imaging evaluation, and serum protein marker test results.

Exclusion Criteria:

* 1. The patient cannot provide a complete and qualified specimen.
* 2. The patient has other primary malignant tumors or serious medical illnesses.
* 3. The patient cannot cooperate with the follow-up.
* 4. Conditions that other researchers deemed inappropriate for continuing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
ctDNA status | Two weeks
  Detect postoperative tissue ctDNA status
ctDNA dynamic detection | 6 months
  ctDNA dynamic monitoring during postoperative adjuvant chemotherapy

SECONDARY OUTCOMES:
Imaging examination | 6 months
  Imaging examination during postoperative adjuvant chemotherapy
Tumor Marker examination | 6 months
  Tumor marker examination during postoperative adjuvant chemotherapy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Francis G, Stein S. Circulating Cell-Free Tumour DNA in the Management of Cancer. Int J Mol Sci. 2015 Jun 19;16(6):14122-42. doi: 10.3390/ijms160614122. PMID 26101870
- [Background] Diehl F, Schmidt K, Choti MA, Romans K, Goodman S, Li M, Thornton K, Agrawal N, Sokoll L, Szabo SA, Kinzler KW, Vogelstein B, Diaz LA Jr. Circulating mutant DNA to assess tumor dynamics. Nat Med. 2008 Sep;14(9):985-90. doi: 10.1038/nm.1789. Epub 2007 Jul 31. PMID 18670422
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348